CLINICAL TRIAL: NCT04047628
Title: A Multicenter Randomized Controlled Trial of Best Available Therapy Versus Autologous Hematopoietic Stem Cell Transplant for Treatment-Resistant Relapsing Multiple Sclerosis (ITN077AI)
Brief Title: Best Available Therapy Versus Autologous Hematopoietic Stem Cell Transplant for Multiple Sclerosis (BEAT-MS)
Acronym: BEAT-MS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Immune Tolerance Network (ITN) (Network); Blood and Marrow Transplant Clinical Trials Network (Network); PPD Development, LP (Industry); Rho Federal Systems Division, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DAIT ITN077AI; UM1AI109565 (NIH); NIAID CRMS ID#: 38573 (Other: DAIT NIAID); BMT CTN 1905 (Other: Bone Marrow and Transplant Clinical Trials Network (BMT CTN))
Record Dates: First submitted 2019-08-05; First posted 2019-08-07 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Relapsing Multiple Sclerosis; Relapsing Remitting Multiple Sclerosis; Secondary Progressive Multiple Sclerosis
Keywords: Treatment-Resistant Relapsing Multiple Sclerosis (MS); Autologous Hematopoietic Stem Cell Transplantation (AHSCT); Autologous Peripheral Blood Stem Cells (PBMCs) Graft; Best Available Therapy (BAT); Disease-Modifying Therapy (DMT); BAT DMT
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis, Chronic Progressive | interventions — Natalizumab; Alemtuzumab; ocrelizumab; Rituximab; Cladribine; ofatumumab; ublituximab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- AHSCT (Experimental): AHSCT: Myeloablative and Immunoablative therapy followed by Autologous Hematopoietic Stem Cell Transplantation
  Participants will undergo:
  1. Mobilization and graft collection: mobilization of peripheral blood stem cells (PBSC) with cyclophosphamide, filgrastim, and dexamethasone. The autologous graft will be collected by leukapheresis and cryopreserved.
  2. Conditioning: high dose myeloablative and immunoablative conditioning with a six-day BEAM chemotherapy and rabbit anti-thymocyte globulin regimen will be initiated ≥30 days after cyclophosphamide mobilization.
  3. Autologous cryopreserved graft infusion: the cryopreserved peripheral blood stem cells (PBSC) graft will be thawed and infused the day following completion of the conditioning regimen. Each bag will be thawed and infused according to institutional standards consistent with the Foundation for the Accreditation of Cellular Therapy (FACT) guidelines. Participants will receive prednisone following graft infusion.
  Interventions: Procedure: Autologous Hematopoietic Stem Cell Transplantation
- Best Available Therapy (BAT) (Active Comparator): Participants randomized to BAT: Best available therapy will be selected by the Site Investigator from: Cladribine (Mavenclad®), natalizumab (Tysabri®), alemtuzumab (Campath®, Lemtrada®), ocrelizumab (Ocrevus®), ublituximab (BRIUMVI™), rituximab (Rituxan®), or ofatumumab (Arzerra®) (after approval by the FDA for relapsing MS).
  Interventions: Biological: Best Available Therapy (BAT)

INTERVENTIONS:
Procedure: Autologous Hematopoietic Stem Cell Transplantation — 1. PBSC mobilization & collection regimen per protocol/ institutional standards includes: intravenous cyclophosphamide (Cytoxan®), 4 grams/m^2); intravenous mesna (Mesnex®),a total delivery of 4 grams/m^2); oral dexamethasone, 10 mg dose, four times daily); subcutaneous filgrastim,10 mcg/kg/day until leukapheresis goal is completed; and CD34+ peripheral blood stem cells collection by leukapheresis.
  2. Conditioning per protocol& institutional standards:
     * 6-day BEAM (e.g. Carmustine (BCNU), Etoposide (VP-16), Cytarbine (Ara-C), and Melphalan) chemotherapy protocol and,
     * rabbit anti-thymocyte globulin (rATG) 2.5 mg/kg/day x2
  3. Autologous cryopreserved graft infusion: The target Cluster of Differentiation (CD)34+ cell dose for infusion is 5 x 10^6 CD34+ cells/kg (minimum 4 x 10^6 CD34+ cells/kg; maximum 7.5 x 10^6 CD34+ cells/kg).
  For 1&2 above: Ideal body weight (IBW) versus Actual Body Weight (ABW) are applicable.
  Other Names: AHSCT
  Arms: AHSCT
Biological: Best Available Therapy (BAT) — Disease-modifying therapy (DMT) selected by the Site Investigator from the below:
  * cladribine
  * natalizumab
  * alemtuzumab
  * ocrelizumab,
  * rituximab,
  * ofatumumab, or
  * ublituximab
  Other Names: natalizumab (Tysabri®); alemtuzumab (Campath®, Lemtrada®); ocrelizumab (Ocrevus®); rituximab (Rituxan®); cladribine (Mavenclad®); ofatumumab (Kesimpta®); ublituximab (BRIUMVI™)
  Arms: Best Available Therapy (BAT)

SUMMARY:
This is a multi-center prospective rater-masked (blinded) randomized controlled trial of 156 participants, comparing the treatment strategy of Autologous Hematopoietic Stem Cell Transplantation (AHSCT) to the treatment strategy of Best Available Therapy (BAT) for treatment-resistant relapsing multiple sclerosis (MS). Participants will be randomized at a 1 to 1 (1:1) ratio.

All participants will be followed for 72 months after randomization (Day 0, Visit 0).

DETAILED DESCRIPTION:
Participant recruitment for this six-year research study focuses on multiple sclerosis (MS) that has remained active despite treatment. This study will compare high dose immunosuppression followed by autologous hematopoietic stem cell transplantation (AHSCT) to best available therapy (BAT) in the treatment of relapsing MS.

MS is a disease caused by one's own immune cells. Normally, immune cells fight infection. In MS, immune cells called T cells, or chemical products made by immune cells, react against the covering or coat (myelin) of nerve fibers in the brain and spinal cord. This leads to stripping the coat from certain nerve fibers (demyelination), and this causes neurologic problems. MS can cause loss of vision, weakness or incoordination, loss or changes in sensation, problems with thinking or memory, problems controlling urination, and other disabilities.

Most individuals with MS first have immune attacks (called relapses) followed by periods of stability. Over time, MS can have episodes of new and worsening symptoms, ranging from mild to disabling. This is called relapsing MS. Relapsing MS includes relapsing remitting MS (RRMS) and secondary progressive MS (SPMS). There are medicines (drugs) to decrease relapses, but these are neither considered to be curative nor, to induce prolonged remissions without continuing therapy.

More than a dozen medicines have been approved for the treatment of relapsing forms of MS. These medicines differ in how safe they are and how well they work. Despite availability of an increasing number of effective medicines, some individuals with relapsing MS do not respond to treatment. Research is being conducted to find other treatments.

High dose immunosuppression followed by autologous hematopoietic stem cell transplantation (AHSCT) has been shown to help relapsing MS in cases where medicines did not work. AHSCT involves collecting stem cells, which are produced in the bone marrow. These stem cells are "mobilized" to leave the bone marrow and move into the blood where they can be collected and stored. Participants will then receive chemotherapy intended to kill immune cells. One's own stored (frozen) stem cells are then given back, through an infusion. This "transplant" of one's stem cells allows the body to form new immune cells in order to restore their immune system. New research suggest that MS might be better controlled with AHSCT than with medicines.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 55 years, inclusive, at the time of the screening Visit -2.
2. Diagnosis of MS according to the 2017 McDonald Criteria139.
3. EDSS ≤ 6.0 at the time of randomization (Day 0).
4. T2 abnormalities on brain MRI that fulfill the 2017 McDonald MRI criteria for dissemination in space139. A detailed MRI report or MRI images must be available for review by the site neurology investigator.
5. Highly active treatment-resistant relapsing MS, defined as ≥ 2 episodes of disease activity in the 36 months prior to the screening visit (Visit -2). The two disease activity episodes will be a clinical MS relapse or MRI evidence of MS disease activity and must meet all the criteria described below:

   1. At least one episode of disease activity must occur following ≥ 1 month of treatment with one of the following: (i) an oral DMT approved by the FDA for the treatment of relapsing MS, or (ii) a monoclonal antibody approved by the FDA for the treatment of relapsing MS, or (iii) rituximab. Qualifying DMTs include: dimethyl fumarate, diroximel fumarate, monomethyl fumarate, teriflunomide, cladribine, daclizumab, ponesimod, siponimod, ozanimod, fingolimod, rituximab, ocrelizumab, natalizumab, alemtuzumab, ublituximab, and ofatumumab, and
   2. At least one episode of disease activity must have occurred within the 12 months prior to the screening visit (Visit -2), and
   3. At least one episode of disease activity must be a clinical MS relapse (see item c.i. below). The other episode(s) must occur at least one month before or after the onset of the clinical MS relapse, and must be either another clinical MS relapse or MRI evidence of disease activity (see item c.ii. below):

   i. Clinical MS relapse must be confirmed by a neurologist's assessment and documented contemporaneously in the medical record. If the clinical MS relapse is not documented in the medical record, it must be approved by the study adjudication committee (see Section 3.5), and ii. MRI evidence of disease activity must include ≥ 1 unique active lesion on one or more brain or spinal cord MRIs. Detailed MRI reports or MRI images must be available for review by the site neurology investigator. A unique active lesion is defined as either of the following:

1. A gadolinium-enhancing lesion, or 2. A new non-enhancing T2 lesion compared to a reference scan obtained not more than 36 months prior to the screening visit (Visit -2).

6. Candidacy for treatment with at least one of the following high efficacy BAT DMTs: cladribine, natalizumab, alemtuzumab, ocrelizumab, ofatumumab, ublituximab and rituximab. Candidacy for treatment for each BAT DMT is defined as meeting all of the following:

1. No prior disease activity episode, as defined in Inclusion Criterion #5, with the candidate BAT DMT, and
2. No contraindication to the candidate BAT DMT, and
3. No treatment with the candidate BAT DMT in the 12 months prior to screening.

   7. Completion of COVID-19 vaccination series, according to the current Centers for Disease Control and Prevention (CDC) Advisory Committee on Immunization Practices (ACIP) recommendations, ≥ 14 days prior to randomization (Day 0).

   8. Positive for VZV antibodies, or completion of at least one dose of the varicella zoster glycoprotein E (gE) Shingrix vaccine at least 4 weeks prior to randomization (Day 0).

   9. Insurance approval for MS treatment with at least one candidate BAT DMT (see Inclusion Criterion #6).

   10. Ability to comply with study procedures and provide informed consent, in the opinion of the investigator.

   11. Females of childbearing potential (defined in Section 5.4.3.1) and males with female partners of childbearing potential are required to adhere to the contraception provisions of Section 5.4.3.1.

   12. For participants who use medicinal or recreational marijuana, willingness to substitute MARINOL® if randomized to AHSCT (Section 5.4.2.6).

Exclusion Criteria:

1. Diagnosis of primary progressive MS according to the 2017 McDonald criteria.
2. History of neuromyelitis optica spectrum disorder or MOG antibody disease.
3. Prior treatment with an investigational agent within 3 months or 5 half-lives, whichever is longer. Agents authorized by the FDA for prevention or treatment of COVID-19 are not considered investigational.
4. Either of the following within one month prior to randomization (Day 0):

   1. Onset of acute MS relapse, or
   2. Treatment with intravenous methylprednisolone 1000 mg/day for 3 days or equivalent.
5. Initiation of any BAT DMT (see Section 5.2.1) between Visit -2 and randomization (Day 0).
6. Brain MRI or cerebrospinal fluid (CSF) examination indicating a diagnosis of progressive multifocal leukoencephalopathy (PML).
7. History of cytopenia consistent with the diagnosis of myelodysplastic syndrome (MDS).
8. Presence of unexplained cytopenia, polycythemia, thrombocythemia or leukocytosis.
9. History of sickle cell anemia or other hemoglobinopathy.
10. Evidence of past or current hepatitis B or hepatitis C infection, including treated hepatitis B or hepatitis C. Hepatitis B surface antibody following hepatitis B immunization is not considered to be evidence of past infection.
11. Presence or history of mild to severe cirrhosis.
12. Hepatic disease with the presence of either of the following:

    1. Total bilirubin ≥ 1.5 times the upper limit of normal (ULN) or total bilirubin ≥ 3.0 times the ULN in the presence of Gilbert's syndrome, or
    2. Alanine Aminotransferase (ALT) or Aspartate Aminotransferase (AST) ≥ 2.0 times the ULN.
13. Positive COVID-19 PCR test, or alternative nucleic acid amplification test (NAAT) per institutional standards, within 14 days prior to randomization (Day 0).
14. Evidence of HIV infection.
15. Positive QuantiFERON - TB Gold,TB Gold Plus, or T-SPOT®.TB test results. PPD tuberculin test may be substituted for QuantiFERON - TB Gold, TB Gold Plus, or T-SPOT®.TB test.
16. Active viral, bacterial, endoparasitic, or opportunistic infections.
17. Active invasive fungal infection.
18. Hospitalization for treatment of infections or parenteral (IV or IM) antibacterials, antivirals, antifungals, or antiparasitic agents within the 30 days prior to randomization (Day 0) unless clearance is obtained from an Infectious Disease specialist.
19. Receipt of live or live-attenuated vaccines within 6 weeks of randomization (Day 0).
20. Presence or history of clinically significant cardiac disease including: a. Arrhythmia requiring treatment with any antiarrhythmia therapy, with the exception of low dose beta blocker for intermittent premature ventricular contractions.

    b. Coronary artery disease with a documented diagnosis of either: i. Chronic exertional angina, or ii. Signs or symptoms of congestive heart failure. c. Evidence of heart valve disease, including any of the following: i. Moderate to severe valve stenosis or insufficiency, or ii. Symptomatic mitral valve prolapse, or iii. Presence of prosthetic mitral or aortic valve.
21. Left ventricular ejection fraction (LVEF) < 50%.
22. Impaired renal function defined as eGFR < 60 mL/min/1.73 m2, according to the CKD-EPI formula144.
23. Forced expiratory volume in one second (FEV1) < 70% predicted (no bronchodilator).
24. Diffusing capacity of the lungs for carbon monoxide (DLCO) (corrected for Hgb) < 70% predicted.
25. Poorly controlled diabetes mellitus, defined as HbA1c > 8%.
26. History of malignancy, except adequately treated localized basal cell or squamous skin cancer, or carcinoma in situ of the cervix. Malignancies for which the participant is judged to be cured will be considered on an individual basis by the study adjudication committee (see Section 3.5).
27. Presence or history of any moderate to severe rheumatologic autoimmune disease requiring treatment, including but not limited to the following: systemic lupus erythematous, systemic sclerosis, rheumatoid arthritis, Sjogren's syndrome, polymyositis, dermatomyositis, mixed connective tissue disease, polymyalgia rheumatica, polychondritis, sarcoidosis, vasculitis syndromes, or unspecified collagen vascular disease.
28. Presence of active peptic ulcer disease, defined as endoscopic or radiologic diagnosis of gastric or duodenal ulcer.
29. Prior history of AHSCT.
30. Prior history of solid organ transplantation.
31. Positive pregnancy test or breastfeeding.
32. Failure to willingly accept or comprehend irreversible sterility as a side effect of therapy.
33. Psychiatric illness, mental deficiency, or cognitive dysfunction severe enough to interfere with compliance or informed consent.
34. History of hypersensitivity to rabbit or Escherichia coli-derived proteins.
35. Any metallic material or electronic device in the body, or other condition that precludes the participant from undergoing MRI with gadolinium administration, as determined by the site radiologist.
36. Presence or history of ischemic cerebrovascular disorders, including but not limited to transient ischemic attack, subarachnoid hemorrhage, cerebral thrombosis, cerebral embolism, or cerebral hemorrhage.
37. Presence or history of other neurological disorders, including but not limited to CNS or spinal cord tumor; metabolic or infectious cause of myelopathy; genetically-inherited progressive CNS disorder; CNS sarcoidosis; or systemic autoimmune disorders potentially causing progressive neurologic disease or affecting ability to perform the study assessments.
38. Presence of any medical comorbidity that the investigator determines will significantly increase the risk of treatment mortality.
39. Presence of any other concomitant medical condition that the investigator deems incompatible with trial participation.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 156 (Estimated)
Dates: Start 2019-12-19 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Multiple Sclerosis (MS) Relapse-Free Survival | From Day 0 (Randomization to Treatment) Up to 36 Months (3 Years)
  MS relapse-free survival, analyzed as time from treatment randomization until MS relapse or death from any cause.

SECONDARY OUTCOMES:
Number of Multiple Sclerosis (MS) Relapses Per Year | From Day 0 (Randomization to Treatment) Up to 72 Months (6 Years)
  Annual Relapse Rate (ARR) time calculated as number of confirmed relapses divided by time in study per year.
The Occurrence of Any Evidence of Multiple Sclerosis (MS) Disease Activity or Death From Any Cause | From Day 0 (Randomization to Treatment) Up to 72 Months (6 Years)
  The occurrence of any evidence of MS disease activity or death from any cause, analyzed as time-to-event.
The Occurence of Confirmed Disability Worsening by the Kurtz Expanded Disability Status Scale (EDSS) | From Day 0 (Randomization to Treatment) Up to 72 Months (6 Years)
  Measured by the Kurtzke Expanded Disability Status Scale performed by the masked (blinded) rater.
  EDSS, defined by:
  * A decrease in EDSS of ≥ 1.0 step(s) compared to the EDSS at randomization (Day 0) and
  * Confirmation of disability improvement ≥ 6 months later. The time of confirmed disability worsening measured by EDSS will be the time of first increase in EDSS ≥ 1.0 step(s).
The Occurrence of Confirmed Disability Improvement by the Kurtz Expanded Disability Status Scale (EDSS) | Day 0 (Randomization to Treatment) Up to Month 72 (6 Years)
  Measured by the Kurtzke Expanded Disability Status Scale performed by the masked (blinded) rater.
  Confirmed disability improvement defined by:
  * A decrease in EDSS of ≥ 1.0 step(s) compared to the EDSS at randomization (Day 0) and
  * Confirmation of disability improvement ≥ 6 months later. The time of confirmed disability improvement measured by EDSS will be the time of first decrease in EDSS ≥ 1.0 step(s).
Whole Brain Volume Change from Pre-Randomization Visit to the follow-up evaluations | From Visit Pre-R Up to 72 Months (6 Years)
  Method of assessment: Magnetic Resonance Imaging (MRI) imaging.
Change in Serum Neurofilament Light Chain (NfL) Concentration | From Day 0 (Randomization to Treatment) Up to 72 Months (6 Years)
  Extent of neurofilament light chain (NfL) concentration in serum is a component of the neuronal cytoskeleton and is released into the cerebrospinal fluid and subsequently blood following neuro-axonal damage.
The Occurrence of Death From Any Cause: All-Cause Mortality | Day 0 (Randomization to Treatment) Up to Month 72 (6 Years)
  Any death, regardless of relationship to treatment.
Proportion of Participants who Experience a Serious Adverse Event (SAE) | From Day 0 (Randomization to Treatment) Up to 72 Months (6 Years)
  An event that results in any of the following outcomes:
  * Death,
  * A life-threatening event that places the participant at immediate risk of death,
  * Inpatient hospitalization or prolongation of existing hospitalization,
  * Persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, or
  * A congenital anomaly or birth defect.
    * Note: Important medical events that may not result in death, be life threatening, or require hospitalization may be considered serious when, based upon appropriate medical judgment, they may jeopardize the participant and may require medical or surgical intervention to prevent one of the outcomes listed in this definition.
  Reference: Code of Federal Regulations Title 21 Part 312.32(a)
Proportion of Participants with a Grade 3 or Higher Infection | From Day 0 (Randomization to Treatment) Up to 72 Months (6 Years)
  In accordance with the criteria set forth in the National Cancer Institute's Common Terminology Criteria for Adverse Events NCI-CTCAE version 5.0, published November 27, 2017.
Proportion of Participants with Progressive Multifocal Leukoencephalopathy (PML) | From Day 0 (Randomization to Treatment) Up to 72 Months (6 Years)
  The occurrence of PML during the course of participation in this study.
  A disease of the white matter of the brain, caused by a virus infection, Polyomavirus JC (JC virus), that targets cells that make myelin--the material that insulates nerve cells (neurons).
Time to Neutrophil Engraftment Among Autologous Hematopoietic Stem Cell Transplantation (AHSCT) Recipients | From Day of Graft Infusion (Receipt of Peripheral Blood Stem Cells-PBSC Infusion) Up to 72 Months (6 Years)
  Neutrophil engraftment is defined as absolute neutrophil count (ANC) > 500/µl on two consecutive measurements on different days.
Proportion of Autologous Hematopoietic Stem Cell Transplantation (AHSCT) Recipients Who Experience Primary or Secondary Graft Failure | From Day of Transplant (Receipt of Peripheral Blood Stem Cells-PBSC Infusion) Up to Day 28 Post Transplant
  Graft failure can either be primary (graft never established) or secondary (loss of an established graft).
  Primary graft failure is the absence of adequate hematopoiesis by Day T28, defined as meeting all of the following conditions:
  * Bone marrow cellularity <5%,
  * Peripheral White Blood Cell Count (WBC) < 500/µl,
  * Peripheral Absolute Neutrophil Count (ANC) < 100/ µl, and
  * Platelets < 10,000/ µl.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey A. Cohen, MD, Study Chair — Mellen Center for MS Treatment and Research, Cleveland Clinic; George E. Georges, MD, Study Chair — Northwestern University; Paolo A. Muraro, MD, PhD, Study Chair — Department of Medicine, Imperial College London
Locations (22):
- United States (22):
  - Stanford Multiple Sclerosis Center, Palo Alto, California
  - Rocky Mountain Multiple Sclerosis Center, University of Colorado School of Medicine, Aurora, Colorado
  - Northwestern University, Evanston, Illinois
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - University of Minnesota Multiple Sclerosis Center, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - John L. Trotter Multiple Sclerosis Center, Washington University School of Medicine in St. Louis, St Louis, Missouri
  - Corinne Goldsmith Dickinson Center for Multiple Sclerosis at Mount Siinai, New York, New York
  - Rochester Multiple Sclerosis Center, University of Rochester, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati (UC) Waddell Center for Multiple Sclerosis, Cincinnati, Ohio
  - Mellen Center for Multiple Sclerosis Treatment and Research, Cleveland Clinic, Cleveland, Ohio
  - Multiple Sclerosis Center, Oregon Health & Science University, Portland, Oregon
  - Penn Comprehensive MS Center, Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Texas Southwestern Medical Center: Division of Multiple Sclerosis and Neuroimmunology, Dallas, Texas
  - Maxine Mesigner Multiple Sclerosis Comprehensive Care Center, Baylor College of Medicine Medical Center, Houston, Texas
  - University of Virginia, Charlottesville, Virginia
  - Virginia Commonwealth University Multiple Sclerosis Treatment and Research Center, Richmond, Virginia
  - Clinical Research Division, Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Multiple Sclerosis Center, Swedish Neuroscience Institute, Seattle, Washington
  - Multiple Sclerosis Center at Northwest Hospital, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Participant level data access and additional relevant materials will be made available upon completion of the trial.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: After completion of the trial, within 24 months status post database lock.
Access Criteria: Registration is available for the Immunology Database and Analysis Portal (ImmPort) at: https://www.immport.org/registration and submit a rationale for the purpose of requesting study data access.
  ImmPort is a long-term archive of clinical and mechanistic data, a National Institute of Allergy and Infectious Diseases Division of Allergy, Immunology and Transplantation (NIAID DAIT)-funded data repository. This archive is in support of the NIH mission to share data with the public. Data shared through ImmPort is provided by NIH-funded programs, other research organizations and individual scientists, ensuring these discoveries will be the foundation of future research.
URL: https://www.immport.org/home

REFERENCES:
- [Background] Nash RA, Hutton GJ, Racke MK, Popat U, Devine SM, Steinmiller KC, Griffith LM, Muraro PA, Openshaw H, Sayre PH, Stuve O, Arnold DL, Wener MH, Georges GE, Wundes A, Kraft GH, Bowen JD. High-dose immunosuppressive therapy and autologous HCT for relapsing-remitting MS. Neurology. 2017 Feb 28;88(9):842-852. doi: 10.1212/WNL.0000000000003660. Epub 2017 Feb 1. PMID 28148635
- [Background] Nash RA, Hutton GJ, Racke MK, Popat U, Devine SM, Griffith LM, Muraro PA, Openshaw H, Sayre PH, Stuve O, Arnold DL, Spychala ME, McConville KC, Harris KM, Phippard D, Georges GE, Wundes A, Kraft GH, Bowen JD. High-dose immunosuppressive therapy and autologous hematopoietic cell transplantation for relapsing-remitting multiple sclerosis (HALT-MS): a 3-year interim report. JAMA Neurol. 2015 Feb;72(2):159-69. doi: 10.1001/jamaneurol.2014.3780. PMID 25546364
- [Background] Cohen JA, Baldassari LE, Atkins HL, Bowen JD, Bredeson C, Carpenter PA, Corboy JR, Freedman MS, Griffith LM, Lowsky R, Majhail NS, Muraro PA, Nash RA, Pasquini MC, Sarantopoulos S, Savani BN, Storek J, Sullivan KM, Georges GE. Autologous Hematopoietic Cell Transplantation for Treatment-Refractory Relapsing Multiple Sclerosis: Position Statement from the American Society for Blood and Marrow Transplantation. Biol Blood Marrow Transplant. 2019 May;25(5):845-854. doi: 10.1016/j.bbmt.2019.02.014. Epub 2019 Feb 19. PMID 30794930
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait
- See also: Immune Tolerance Network (ITN) — http://www.immunetolerance.org
- See also: Visit this ITN Study website for more information — http://beat-ms.org/